CLINICAL TRIAL: NCT01574638
Title: Phase I Clinical Trial of the Pharmacokinetics of High-dose Daily Rifapentine, Given as a Single Dose or in Divided Doses to Healthy Volunteers
Brief Title: Evaluating the Pharmacokinetics of High-Dose Rifapentine When Given as a Single Dose or in Divided Doses to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5311; 11859 (Registry Identifier: DAIDS ES); ACTG5311; ACTG 5311
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2015-10

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1B (Experimental): Participants in Arm 1B will receive RPT based on weight at entry, at a dose of 20 mg/kg once daily with a low-fat breakfast, on Days 1 to 14. Participants will not receive RPT on Days 15 to 42 and will resume receipt of RPT on Days 43 to 56, at a dose of 10 mg/kg twice daily with low-fat meals.
  Interventions: Drug: Rifapentine (RPT)
- Arm 1A (Experimental): Participants in Arm 1A will receive RPT based on weight at entry, at a dose of 10 mg/kg twice daily with low-fat meals, on Days 1 to 14. Participants will not receive RPT on Days 15 to 42 and will resume receipt of RPT on Days 43 to 56, at a dose of 20 mg/kg once daily with a low-fat breakfast.
  Interventions: Drug: Rifapentine (RPT)
- Arm 2A (Experimental): Participants in Arm 2A will receive RPT based on weight at entry, at a dose of 15 mg/kg once daily with a boiled egg, on Days 1 to 14. Participants will not receive RPT on Days 15 to 42 and will resume receipt of RPT on Days 43 to 70, at a dose of 15 mg/kg once daily with a low-fat breakfast.
  Interventions: Drug: Rifapentine (RPT)
- Arm 2B (Experimental): Participants in Arm 2B will receive RPT based on weight at entry, at a dose of 15 mg/kg once daily with a low-fat breakfast, on Days 1 to 14. Participants will not receive RPT on Days 15 to 42 and will resume receipt of RPT on Days 43 to 56, at a dose of 15 mg/kg once daily with a boiled egg.
  Interventions: Drug: Rifapentine (RPT)

INTERVENTIONS:
Drug: Rifapentine (RPT) — Participants will receive 150-mg RPT tablets orally either once or twice daily, with total tablet number/dosage amount varying according to weight at entry and arm assignment and following dosing tables in the protocol.

SUMMARY:
This study will evaluate two different ways to give rifapentine (RPT), a drug that may help shorten treatment duration for tuberculosis (TB) disease.

DETAILED DESCRIPTION:
TB continues to be a major global health problem, with an estimated 9.4 million new cases and 1.3 million deaths from TB in 2009. Effective treatment is available, but the current standard therapy consists of 4 different drugs that must be given for 6 months to be effective. RPT is a rifamycin antibiotic approved by the Food and Drug Administration (FDA) to be given twice weekly during the intensive phase of TB treatment and once weekly during the continuation phase of TB treatment. However, studies using this regimen have seen high relapse rates of TB; use of higher and/or more frequent doses may be necessary to attain higher cure rates. This study will evaluate 2 strategies for optimizing RPT exposure: dividing the daily dose in order to increase absorption/overall drug exposure and providing the dose together with food.

Participants will be randomly assigned to one of 4 arms: Arm 1A, Arm 1B, Arm 2A, or Arm 2B. The first 12 participants who indicate that they are willing to remain on the study for up to 12 weeks will be assigned to Arm 2A; all others will be randomized to Arm 1A, 1B, or 2B. Participants in all arms will receive daily RPT from Day 1 to 14, followed by a washout period from Day 15 to 42 during which no RPT will be given, followed by a second period of daily RPT from Day 43 to 56 (and continuing through Day 70 for participants in Arm 2A). Arms 1A and 2B will evaluate twice-daily versus once-daily RPT taken with low-fat meals; Arms 2A and 2B will evaluate once-daily RPT given with an egg versus with a low-fat breakfast.

Total study duration will range from 63 to 70 days for Arms 1A, 1B, and 2B, with 10 study visits: 4 intensive pharmacokinetic (PK) sampling visits (at Days 0 to 2, 13 to 15, 42 to 44, and 55 to 57) and 6 other visits at screening and Days 7, 21, 35, and 49, with the final visit between Days 63 and 70. Total study duration for Arm 2A will range from 77 to 84 days, with 12 study visits: 5 intensive PK sampling visits (over Days 0 to 2, 13 to 15, 42 to 44, 55 to 57, and 69 to 71) and 7 other visits at screening and Days 7, 21, 35, 49, and 64, with the final visit between Days 77 and 84. Intensive PK visits will require the participant to be admitted to the clinic for 1 or 2 nights and to have blood collected multiple times. Interim study visits may consist of giving a medical history, undergoing a physical exam and blood collection, and undergoing a pregnancy test for women of reproductive potential. Participants also will be required to keep a diary of the times they took outpatient study drugs, any medications taken other than the study drug, and any symptoms experienced.

ELIGIBILITY:
Inclusion Criteria:

* Weight of 50 to 100 kg, inclusive
* Absence of HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit within 21 days prior to study entry. NOTE: The term "licensed" refers to a U.S. FDA-approved kit.
* Females of reproductive potential (defined as women who have not been postmenopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, and do not have documentation of having undergone a sterilization procedure [e.g., hysterectomy or bilateral oophorectomy or salpingectomy]) must have a negative serum or urine beta-human choriogonadotropin (β-HCG) pregnancy test performed within 48 hours prior to entry. The urine test must have a sensitivity of at least 25 mlU/mL and be performed at a laboratory with Clinical Laboratory Improvement Amendment (CLIA) certification or its equivalent.

  * If participating in sexual activity that could lead to pregnancy, females must agree to use at least one reliable form of contraceptive while receiving the protocol-specified medications and for 1 week after stopping study medications. At least one (but preferably two) of the following contraceptives MUST be used appropriately:
  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)

    * NOTE: Hormone-based contraceptives are contraindicated with RPT and therefore may not be used as a form of contraception during this study.
* Ability and willingness of volunteer to provide written informed consent
* Laboratory values obtained within 21 days prior to entry:

  * Serum alanine aminotransferase (ALT) less than or equal to 1.2 times the upper limit of normal (ULN)
  * Total bilirubin level less than or equal to 1.2 times the ULN
  * Serum creatinine less than or equal to 1.5 mg/dL
  * Hemoglobin greater than or equal to 12.0 g/dL for men, greater than or equal to 11.0 g/dL for women
  * Platelet count greater than or equal to 125,000/mm^3
  * Absolute neutrophil count greater than or equal to 1,250/mm^3
  * Serum albumin greater than or equal to 3.5 g/dL
  * Hepatitis C antibody negative

Exclusion Criteria:

* Breastfeeding
* Within 30 days prior to entry, use of any prescription medication known to inhibit or induce cytochrome P (CYP)3A metabolizing enzymes (refer to the manufacturers' package inserts for individual drugs). See list posted on the A5311 protocol-specific webpage (PSWP).
* Known intolerance of or allergy to chicken eggs
* Use of rifamycin antibiotics within 60 days prior to entry
* Planned use during the study of prescription medications, herbal supplements, nutritional supplements, or over-the-counter medications except as follows: multivitamins, acetaminophen (up to 650 mg every 6 hours as an analgesic), ibuprofen (up to 600 mg twice daily), naproxen (up to 500 mg twice daily for pain or headache), and Benadryl (diphenhydramine, up to 25 mg daily for insomnia or seasonal allergies) are permitted. The use of topical or locally-acting drugs (e.g., eye drops, IUDs, skin ointments) will be considered on a case-by-case basis.
* Within 14 days prior to study entry, hospitalization for any reason or pharmacotherapy for serious illness
* Within 14 days prior to study entry, use of any prescription medication(s)
* Receipt of any investigational study drug within 21 days prior to study entry
* Known allergy/sensitivity or any hypersensitivity to rifamycins, including rifampin, rifabutin, and rifapentine
* Presence of any condition interfering with normal gastrointestinal anatomy or motility that could interfere with drug absorption or excretion (including cholecystectomy, peptic ulceration, inflammatory bowel disease, or pancreatitis)
* History or evidence of clinically significant (as determined by site investigator) cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, or immunologic disease(s)
* Any medical condition that, in the opinion of the site investigator, would interfere with the participant's ability to participate in the study
* Active illicit drug use or dependence or alcohol dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* History of TB infection or site investigator suspicion of current active TB
* Inability to abstain from grapefruit and grapefruit juice for the duration of the study
* Inability to adhere to the dietary requirements of the study (e.g., low-fat meal or boiled egg prior to drug doses during the study drug administration periods)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
RPT PK parameter: area under the curve over 24 hours (AUC 0 to 24h) | Measured at Days 14 and 56
  Measured in Group 1, when given at a dose of 20 mg/kg once daily (Arm 1B) and when given at a dose of 10 mg/kg twice daily (Arm 1A)
RPT PK parameter: AUC 0 to 24h | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
Grade 2 or higher signs and symptoms observed while on study beginning with the first dose of study drug and continuing through the follow-up period | Measured through Day 84

SECONDARY OUTCOMES:
RPT PK parameter: maximum observed plasma concentrations (Cmax) | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
Cmin (trough) values | Measured at Days 1, 7, 14, 43, 49, 56, 64, and 70
Metabolizer status of human genetic variants/polymorphisms in gene SLCO1B1 and possibly other genes that are thought to affect PK of RIF | Measured at Day 0
RPT PK parameter: minimum observed plasma concentration (Cmin) | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT PK parameter: oral clearance (CL/F) | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT PK parameter: elimination half-life (T 1/2) | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT metabolite desacetyl-rifapentine (desRPT) PK parameter: AUC 0 to 24h | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT metabolite desRPT PK parameter: Cmax | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT metabolite desRPT PK parameter: Cmin | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT metabolite desRPT PK parameter: CL/F | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT metabolite desRPT PK parameter: T1/2 | Measured at Days 14 and 56
  Measured in Group 1, when RPT is given at a dose of 20 mg/kg once daily (Arm 1B) and at a dose of 10 mg/kg twice daily (Arm 1A)
RPT PK parameter: Cmax | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT PK parameter: Cmin | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT PK parameter: CL/F | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT PK parameter: T1/2 | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT metabolite desRPT PK parameter: AUC 0 to 24h | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT metabolite desRPT PK parameter: Cmax | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT metabolite desRPT PK parameter: Cmin | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT metabolite desRPT PK parameter: CL/F | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT metabolite desRPT PK parameter: T1/2 | Measured at Days 14 and 56
  Measured in Group 2, when RPT is given at a dose of 15 mg/kg once daily with a boiled egg (Arm 2A) and at a dose of 15 mg/kg once daily with a low-fat meal (Arm 2B)
RPT and its metabolite desRPT PK parameter AUC 0 to 24h at steady state when given at a dose of 20 mg/kg once daily (Group 1) and at a dose of 15 mg/kg once daily (Group 2 ) | Measured at Days 1, 14, 43, 56, and 70
RPT and its metabolite desRPT PK parameter Cmax at steady state when given at a dose of 20 mg/kg once daily (Group 1) and at a dose of 15 mg/kg once daily (Group 2 ) | Measured at Days 1, 14, 43, 56, and 70
RPT and its metabolite desRPT PK parameter Cmin at steady state when given at a dose of 20 mg/kg once daily (Group 1) and at a dose of 15 mg/kg once daily (Group 2 ) | Measured at Days 1, 14, 43, 56, and 70
RPT and its metabolite desRPT PK parameter CL/F at steady state when given at a dose of 20 mg/kg once daily (Group 1) and at a dose of 15 mg/kg once daily (Group 2 ) | Measured at Days 1, 14, 43, 56, and 70
RPT and its metabolite desRPT PK parameter T1/2 at steady state when given at a dose of 20 mg/kg once daily (Group 1) and at a dose of 15 mg/kg once daily (Group 2 ) | Measured at Days 1, 14, 43, 56, and 70
RPT and its metabolite desRPT PK parameter area under the curve extrapolated to infinity (AUC 0 to inf) | Measured after single dose on Days 1 and 43
RPT and its metabolite desRPT PK parameter CL/F | Measured after single dose on Days 1 and 43
RPT and its metabolite desRPT PK parameter T1/2 | Measured after single dose on Days 1 and 43
RPT and its metabolite desRPT PK parameter AUC 0 to 24h | Measured after multiple dose on Days 14 and 56
RPT and its metabolite desRPT PK parameter CL/F | Measured after multiple dose on Days 14 and 56
RPT and its metabolite desRPT PK parameter T1/2 | Measured after multiple dose on Days 14 and 56

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee

REFERENCES:
- [Background] Zvada SP, Van Der Walt JS, Smith PJ, Fourie PB, Roscigno G, Mitchison D, Simonsson US, McIlleron HM. Effects of four different meal types on the population pharmacokinetics of single-dose rifapentine in healthy male volunteers. Antimicrob Agents Chemother. 2010 Aug;54(8):3390-4. doi: 10.1128/AAC.00345-10. Epub 2010 Jun 1. PMID 20516273
- [Background] Benator D, Bhattacharya M, Bozeman L, Burman W, Cantazaro A, Chaisson R, Gordin F, Horsburgh CR, Horton J, Khan A, Lahart C, Metchock B, Pachucki C, Stanton L, Vernon A, Villarino ME, Wang YC, Weiner M, Weis S; Tuberculosis Trials Consortium. Rifapentine and isoniazid once a week versus rifampicin and isoniazid twice a week for treatment of drug-susceptible pulmonary tuberculosis in HIV-negative patients: a randomised clinical trial. Lancet. 2002 Aug 17;360(9332):528-34. doi: 10.1016/s0140-6736(02)09742-8. PMID 12241657
- [Derived] Dooley KE, Savic RM, Park JG, Cramer Y, Hafner R, Hogg E, Janik J, Marzinke MA, Patterson K, Benson CA, Hovind L, Dorman SE, Haas DW; ACTG A5311 Study Team. Novel dosing strategies increase exposures of the potent antituberculosis drug rifapentine but are poorly tolerated in healthy volunteers. Antimicrob Agents Chemother. 2015;59(6):3399-405. doi: 10.1128/AAC.05128-14. Epub 2015 Mar 30. PMID 25824215